CLINICAL TRIAL: NCT00137059
Title: Acetaminophen-induced Hepatotoxicity in Chronic Alcohol Abusers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Marco L.A. Sivilotti (Other)
Responsible Party: Sponsor-Investigator, Dr. Marco L.A. Sivilotti, Professor of Emergency Medicine, and of Biomedical & Molecular Science, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PSI R02-52
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hepatotoxicity

INTERVENTIONS:
Drug: acetaminophen sustained-release

SUMMARY:
It is widely believed that people who abuse alcohol can sustain a liver injury after taking doses of acetaminophen just above the recommended maximum dose. This study is designed to look at the interaction between acetaminophen, liver injury and alcohol abuse. Subjects will undergo baseline tests to ensure that they do not have liver damage at the time of enrollment. Each subject will be randomly assigned to receive either a therapeutic dose of acetaminophen or a placebo three times a day for four days. Subjects will have blood work drawn on a daily basis to monitor the status of the liver. These tests will include conventional markers of liver injury in addition to a novel biomarker of liver function, a-GST. Previous work in the investigators' group has shown that a-GST is a more sensitive indicator of liver injury following acetaminophen overdose (Sivilotti 1999, Sivilotti 2002 x 2). However, it has never been used to study the alcoholic population. The investigators believe that a-GST may detect a subclinical acetaminophen-induced liver injury that has previously gone unrecognized in the alcoholic population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who self-report consuming at least 6 drinks per day, daily, for at least 6 weeks and who are currently enrolled at the Detoxification Center, Hotel Dieu Hospital.
* Last alcohol consumption occurring between 12 and 72 hours prior to screening for study.

Exclusion Criteria:

* Individuals with a self-reported or previously documented history of hepatitis A, B, C or HIV.
* Individuals who have ingested any acetaminophen regardless of dose in the previous 48 hours.
* Individuals who have ingested > 4 grams of acetaminophen/day in any of the previous 7 days.
* Individuals < 18 years of age.
* Individuals with abnormal liver function at baseline (defined as AST or ALT > 120 IU/L, International Normalized Ratio [INR] > 1.5, and a-GST > 7.5 7 :g/L).
* Individuals who have an allergy or sensitivity to acetaminophen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-11; Study Completion 2005-05

PRIMARY OUTCOMES:
serum a-GST relative to baseline

SECONDARY OUTCOMES:
conventional liver function tests (LFTs)

CONTACTS AND LOCATIONS:
Overall Officials: Marco LA Sivilotti, MD, MSc, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Bartels S, Sivilotti M, Crosby D, Richard J. Are recommended doses of acetaminophen hepatotoxic for recently abstinent alcoholics? A randomized trial. Clin Toxicol (Phila). 2008 Mar;46(3):243-9. doi: 10.1080/15563650701447020. PMID 18344107